CLINICAL TRIAL: NCT06038617
Title: A Prospective, Randomized, Open-label Clinical Trial to Assess the Safety of Simultaneous Vaccination With mRNA COVID-19 Vaccine and Other Vaccines in Young Children Aged 6 Months to <5 Years.
Brief Title: Safety of Simultaneous mRNA COVID-19 Vaccine With Other Childhood Vaccines in Young Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Kaiser Permanente (Other); Columbia University (Other); Children's Hospital Medical Center, Cincinnati (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00113014
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-06

CONDITIONS: Fever After Vaccination; Fever; Seizures Fever
Keywords: COVID vaccine; Fever following vaccination
MeSH Terms: conditions — Fever; Seizures, Febrile | interventions — CVnCoV COVID-19 vaccine; BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273; measles, mumps, rubella, varicella vaccine; Hepatitis A Vaccines; Hepatitis B Vaccines; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Simultaneous vaccination arm (Experimental): The simultaneous vaccination group will receive routine childhood vaccinations and mRNA COVID-19 vaccination at Visit 1, followed by a health education visit without vaccination at Visit 2.
  Interventions: Biological: mRNA COVID-19 Vaccine; Biological: Routine Childhood Vaccinations
- Sequential vaccination arm (Experimental): The sequential vaccination group will receive routine childhood vaccinations at Visit 1, followed by a health education visit with mRNA COVID-19 vaccination at Visit 2.
  Interventions: Biological: mRNA COVID-19 Vaccine; Biological: Routine Childhood Vaccinations

INTERVENTIONS:
Biological: mRNA COVID-19 Vaccine — ACIP Recommended Vaccine
  Other Names: Pfizer COVID-19 Vaccine, Moderna COVID-19 Vaccine
Biological: Routine Childhood Vaccinations — ACIP Recommended Vaccines
  Other Names: Pneumococcal, DTaP, Haemophilus Influenzae Type B, MMR, Varicella, MMRV, Hepatitis A, Inactivated Poliovirus, Hepatitis B, Rotavirus, Influenza vaccines

SUMMARY:
This is a prospective, randomized, open-label clinical trial to evaluate the safety of COVID-19 vaccination and other routine childhood vaccines given simultaneously at Visit 1, as compared to sequential vaccination of COVID-19 vaccine and other vaccines at separate visits (Visits 1 and 2).

DETAILED DESCRIPTION:
Parent(s) or legal authorized representative(s) (LAR) will assess fever and other solicited systemic adverse events on the day of vaccination (Day 1) and the next 6 days (through Day 7) following Visit 1 and Visit 2 using either a web-based data collection system or a paper memory aid. Serious adverse events and adverse events of special interest will be captured during the entire study period. Parental/LAR perceptions about their child's vaccine schedule will be assessed on Day 7 following Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Child 6 months through <5 years of age at time of enrollment.
* Child is due to receive mRNA COVID-19 vaccine and at least one other routinely recommended non-live vaccine per CDC or ACIP recommendations.
* Parental/LAR intention of child receiving mRNA COVID-19 vaccine and at least one recommended non-live vaccine.
* The parent/LAR must be willing and capable of providing permission for their child to participate through the written informed consent process.
* The parent/LAR must be available for follow-up and must at minimum have telephone access.
* The parent/LAR must agree to sign a medical release for the child so that study personnel may obtain medical information about the child's health (if needed).
* The parent/LAR must be willing to delay COVID-19 vaccination for their child for up to 3 weeks.
* The parent/LAR must be able to read English or Spanish.

Exclusion Criteria:

* History of any seizure (including febrile seizure) or first degree relative (biologic parent or biologic sibling including half-sibling) with a history of febrile seizure.
* Contraindication to mRNA COVID-19 vaccine: A history of a severe allergic reaction (e.g., anaphylaxis) after a previous dose or to a component of the COVID-19 vaccine or a known diagnosed allergy to a component of COVID-19 vaccine.
* A history of a severe allergic reaction (e.g., anaphylaxis) after a previous dose or to a component of a vaccine administered on the day of study enrollment.
* For children receiving DTaP vaccine (alone or combination vaccine): Encephalopathy (e.g., coma, decreased level of consciousness, prolonged seizures), not attributable to another identifiable cause, within 7 days of administration of previous dose of DTP or DTaP.
* Received any other non-live vaccines within 14 days prior to enrollment or any other live vaccines within 28 days prior to enrollment.
* Intention to receive non-COVID-19 non-live or live vaccines during the 4 weeks after Visit 1; vaccines may be administered after enrollment if deemed a personal or public health priority by the health care provider caring for this patient or the study team.
* Received prior COVID-19 vaccine as part of a clinical trial.
* Received any experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) within 28 days prior to enrollment in this study or expects to receive an experimental/investigational agent during the study.
* A moderate to severe acute illness and/or a reported temperature ≥ 100.4°F (≥38.0°C) within 48 hours prior to enrollment or a temperature (measured by temporal artery thermometer) ≥100.4°F (≥38.0°C) at the time of enrollment. (This may result in a temporary delay of vaccination).
* Receipt of an antipyretic medication (acetaminophen or ibuprofen) within 72 hours prior to enrollment (this may result in a temporary delay of vaccination) or planned receipt of a prophylactic antipyretic medication on the day of and/or days following vaccination prior to any measured increase in temperature in anticipation of a fever (this exclusion does not apply if the Parent/LAR indicates they might administer antipyretics or analgesics after vaccination to reduce a fever or pain).
* Immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy since birth.
* Long term (at least 14 days of prednisone 2 mg/kg/day or equivalent other glucocorticoid) use of any parenteral steroids or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the 6 months prior to enrollment (topical and nasal steroids are allowed).
* Has an active case of COVID-19 infection.
* History of multisystem inflammatory syndrome (MIS-C).
* History of myocarditis or pericarditis.
* Has any condition that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.
* Any child or grandchild of a study investigator or study team member.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 344 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Fever Following Vaccination | 2 Days Post-Administration
  Number of children with fever (temperature ≥ 38.0°C or ≥ 100.4°F) on day 1 and/or day 2 following Visit 1 and/or Visit 2.

SECONDARY OUTCOMES:
Number of Participants with Fever Following Visit 1 | 2 Days Post Administration
  Number of children with fever (temperature ≥ 38.0°C or ≥ 100.4°F) on day 1 and/or day 2 following Visit 1
Number of Participants with Fever Following Visit 2 | 2 Days Post Administration
  Number of children with fever (temperature ≥ 38.0°C or ≥ 100.4°F) on day 1 and/or day 2 following Visit 2
Number of Participants with Grade 2 and/or 3 Fever Following Visit 1 | 2 Days Post Administration
  Number of children with moderate/severe fever (Grade 2 and/or 3) on day 1 and/or day 2 following Visit 1. (Moderate/severe fever: ≥ 38.4°C or ≥ 101.2°F)
Number of Participants with Grade 2 and/or 3 Fever Following Visit 2 | 2 Days Post Administration
  Number of children with moderate/severe fever (Grade 2 and/or 3) on day 1 and/or day 2 following Visit 2. (Moderate/severe fever: ≥ 38.4°C or ≥ 101.2°F)
Number of Participants with Grade 2 and/or 3 Fever Following Visit 1 and Visit 2 Combined | 2 Days Post Administration
  Number of children with moderate/severe fever (Grade 2 and/or 3) on day 1 and/or day 2 following Visit 1 and Visit 2 combined. (Moderate/severe fever: ≥ 38.4°C or ≥ 101.2°F)
Number of Participants with Medical Care Utilization - Visit 1 | 2 Days Post Administration
  Number of children with medical care utilization (medical advice (telephone, patient portal),urgent care visit, emergency department visit, and hospital admission) for fever on day 1 and/or day 2 following Visit 1.
Number of Participants with Medical Care Utilization - Visit 2 | 2 Days Post Administration
  Number of children with medical care utilization (medical advice (telephone, patient portal),urgent care visit, emergency department visit, and hospital admission) for fever on day 1 and/or day 2 following Visit 2.
Number of Participants with Medical Care Utilization - Visit 1 and Visit 2 Combined | 2 Days Post Administration
  Number of children with medical care utilization (medical advice (telephone, patient portal), urgent care visit, emergency department visit, and hospital admission) for fever on day 1 and /or day 2 following Visit 1 and Visit 2 combined.
Number of Participants who Received Antipyretics - Visit 1 | 2 Days Post Administration
  Number of children who received antipyretics on day 1 and/or day 2 following Visit 1.
Number of Participants who Received Antipyretics - Visit 2 | 2 Days Post Administration
  Number of children who received antipyretics on day 1 and/or day 2 following Visit 2.
Number of Participants who Received Antipyretics - Visit 1 and Visit 2 Combined | 2 Days Post Administration
  Number of children who received antipyretics on day 1 and/or day 2 following Visit 1 and Visit 2 combined.
Number of Participants with Defined Systemic Reactogenicity Events | Up to 7 Days Post Administration
  Tables summarizing each solicited local and systemic reactogenicity event by maximum classification (none, mild, moderate, and severe), as well as by moderate or severe
The Number and Percent of Individuals with At Least One Serious Adverse Event | Up to 105 Days Post Administration
  The number and percent of serious adverse events observed and description of each event

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Smith, MD, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - Kaiser Permanente Northern California, Oakland, California
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT06038617/ICF_000.pdf